CLINICAL TRIAL: NCT06319222
Title: Implementation of a Digital Clinic for Alcohol-associated Liver Disease and Alcohol Use Disorder (DALC): A Randomized Pragmatic Clinical Trial
Brief Title: Implementation of a Digital Clinic for Alcohol-associated Liver Disease and Alcohol Use Disorder (DALC)
Acronym: DALC
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: Ria Health (Industry)
Responsible Party: Principal Investigator, Douglas (Doug) A. Simonetto, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 23-007870
Record Dates: First submitted 2024-03-13; First posted 2024-03-19 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-05

CONDITIONS: Alcohol Use Disorder; Liver Diseases
Keywords: Alcohol; Liver; Disorder
MeSH Terms: conditions — Alcoholism; Liver Diseases; Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard of Care Arm (No Intervention): Primary care providers will treat subject per standard of care utilizing the Interactive Care Plan program.
- Digital Clinic Arm (Other): The Ria Treatment Platform (RTP) application will be downloaded onto the patient's smart phone or tablet.
  Interventions: Other: DALC Digital Clinic

INTERVENTIONS:
Other: DALC Digital Clinic — Providers randomized to the intervention arm will be able to refer their patients with ALD, to the DALC in addition to standard of care. Patients with providers randomized to the intervention arm will be consented by the study team. After appropriate consent, the referred patients will be instructed by our study team to download the RTP application in their smart devices (smartphones or tablets).
  Arms: Digital Clinic Arm

SUMMARY:
The purpose of this study is to determine whether a multidisciplinary digital clinic will improve health outcomes, reduce costs, increase access, and improve provider satisfaction.

The primary aim of this study is to improve clinical outcomes in patients with ALD through the implementation of a novel digital health platform for personalized multi-disciplinary treatment of patients with ALD and AUD. Secondary aims include improvement in provider and patient-reported outcomes including satisfaction with AUD treatment.

DETAILED DESCRIPTION:
This will be a pilot study with a pragmatic trial design wherein all hepatology providers at the Mayo Clinic in Rochester, MN and Scottsdale, AZ will be invited to participate in the study. Consented providers will be randomized to the Digital ALD/AUD Clinic (DALC) arm or standard of care. Provides randomized to standard of care arm will continue to enroll their patients with ALD in the Interactive Care Plan (ICP), a nursing led program started at Mayo in 2021 for longitudinal remote care of patients with compensated and decompensated cirrhosis. All patients will receive nursing education on alcohol abstinence at ICP enrollment and longitudinal management of their liver disease (current state). Providers randomized to the intervention arm will be able to refer their patients with ALD, to the DALC in addition to standard of care.

The target sample size will be 40 providers (20 providers per arm) and the investigators anticipate 150 patients with ALD will be seen during the study period across both arms. The number of ICP eligible patients seen versus the number of ICP referred patients will be recorded for all providers. Clinically relevant outcomes including hepatic decompensation, MELD 3.0 score, liver chemistries, alcohol use or relapse, liver-related hospitalizations, medication compliance, and mortality will be recorded as part of current ICP program, in both arms. Data will be collected retrospectively from the available medical records at the end of the study period, and no research contact will be made with the patients after initial consent for those patients being offered the DALC. The study duration will be 6 months after the initial Hepatology appointment. At study enrollment and completion, providers will be asked to fill out a survey regarding their satisfaction with ALD/AUD treatment. Consented providers will be informed that they may drop out of the study at any time.

ELIGIBILITY:
Inclusion Criteria:

* Provider-Hepatology Providers at Mayo Clinic Rochester and Scottsdale
* Patient-Age ≥ 18 y.o.
* Patient-Alcohol-associated liver disease

Exclusion Criteria:

* Provider-Providers in other divisions
* Patient-Inability to provide consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-03-12 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Median delta MELD-3.0 from baseline to end of study. | 6 months
  The primary aim of this study is to improve clinical outcomes in patients with ALD as defined as median delta MELD-3.0 from baseline to the end of the study.

SECONDARY OUTCOMES:
Sustained alcohol abstinence | 6 months
  Secondary aims include sustained alcohol abstinence which is obtained by asking the patient if they are continuing to not drink alcohol
Reduction of Number of hospitalizations | 6 months
  Secondary outcome measures include a reduction of number of hospitalizations in the DALC arm compared to the standard of care arm.
Greater provider satisfaction in DALC arm | 6 months
  Secondary outcome measures include greater provider satisfaction with AUD management in the DALC compared to standard of care based on surveys answered by providers. Provider outcome will be assessed by providing the provider a 12 question questionnaire with options to answer Extremely satisfied (5 pts), moderately satisfied (4 pts), neutral (3 pts), moderately dissatisfied (2 pts), very dissatisfied (1pt). The greater the points the greater the satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Douglas Simonetto, MD, Principal Investigator — Mayo Clinic
Locations (2):
- United States (2):
  - Mayo Clinic Arizona, Scottsdale, Arizona
  - Mayo Clinic, Rochester, Minnesota

IPD SHARING:
Plan to Share IPD: No